CLINICAL TRIAL: NCT07282327
Title: The Efficacy and Safety of Female Autologous Platelet-Rich Plasma (PRP) Co-incubation With Husband's Sperm in the Intrauterine Insemination (IUI) to Improve Clinical Pregnancy Rate: A Prospective, Randomized Controlled Trial.
Brief Title: Female Autologous Platelet-Rich Plasma (PRP) Co-incubation With Husband's Sperm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025.450-T
Record Dates: First submitted 2025-08-12; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Reproductive Issues

STUDY DESIGN:
Intervention Model Description: (i) intervention group: female PRP co-incubation with husband's sperm in the IUI (ii) control group: non-PRP in the conventional IUI.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Control group (non-PRP in the conventional IUI)
  Interventions: Other: Sham Comparator: Control group
- Intervention group (Experimental): Intervention group (Female PRP co-incubation with husband's sperm in the IUI)
  Interventions: Other: Female PRP co-incubation with husband's sperm in the IUI

INTERVENTIONS:
Other: Female PRP co-incubation with husband's sperm in the IUI — Intervention group (Female PRP co-incubation with husband's sperm in the IUI)
  Arms: Intervention group
Other: Sham Comparator: Control group — Control group (non-PRP in the conventional IUI)
  Arms: Control group

SUMMARY:
Hypotheses:

We hypothesize that infertility patients undergoing IUI who receive female autologous platelet-rich plasma (PRP) co-incubation with husband's sperm would have higher clinical pregnancy rate.

Aims:

* To determine if the use of female autologous platelet-rich plasma (PRP) co-incubation with husband's sperm in the IUI will show higher clinical pregnancy rate (CPR). Clinical pregnancy rate as determined by a positive serum beta-hCG test result and at least one gestational sac at 6 weeks gestation
* To assess the safety of female PRP co-incubation with husband's sperm in the IUI.

Primary outcome:

To compare the incidence of clinical pregnancy outcome in those infertility patients undergoing IUI with female PRP co-incubation with husband's sperm group and non-PRP group.

Secondary outcomes:

* To evaluate the safeness between the female PRP co-incubation with husband's sperm in the IUI group and non-PRP group, including potential infection rate or other complications such as ectopic pregnancy and molar pregnancy
* To evaluate the sperm quality between the intervention group and control group

Data analysis: Data analysis will be performed using Statistical Packages of Social Sciences for Windows

Expected results: The investigators expect that a 50% pregnancy rate increase after the application of female PRP co-incubation with husband's sperm in the IUI

DETAILED DESCRIPTION:
Outcome measures

Primary outcome:

To measure the rate of clinical pregnancy outcome in subjects undergoing IUI with PRP co-incubation with husband's sperm group than non-PRP group. Clinical pregnancy rate as determined by a positive serum beta-hCG test result at 6 weeks gestation and ultrasound scanning will be performed to confirm at least one gestational sac around 2 to 3 months after IUI.

Secondary outcomes:

* To evaluate the rate of potential infection or other complications such as ectopic pregnancy and molar pregnancy in the intervention group and control group
* Assessment of sperm quality Sperm quality will be assessed before raw semen, post isolated processed semen and after female PRP co-incubation with the processed semen

Sample size IUI's average clinical pregnancy rate is 10.1% in the past five years at Assisted Reproductive Technology Unit of the department of Obstetrics and Gynecological in the Prince of Wales Hospital, we assume a 50% pregnancy rate increase after the application of female PRP co-incubation with husband's sperm in the IUI, the pregnancy rate is expected to be 15.15% in the sample size estimation. With power calculations (G*Power3.1.9.7; t tests-Means: difference of two independent means), 64 couples (128 patients) in each arm would provide a two-sided 80% power with an alpha of 0.05. We aim to recruit a total of 144 couples (288 patients), that is 72 couples (144 patients) in each arm, to account for a 10% dropout rate.

Subjects undergoing IUI will be included in the study if they fulfilled the inclusion criteria. The consented subjects will be randomized into two groups via simple random sampling. The subjects' names will be drawn randomly from a pool in which each had an equal probability of being chosen.

* Intervention group (Female PRP co-incubation with husband's sperm in the IUI)
* Control group (non-PRP in the conventional IUI)

Data processing and analysis The researchers will ensure the confidentiality of sensitive data by minimizing the number of personnel who handles subject data. The computer data will be encrypted as required to maximize security. All paper documents will be locked in filing cabinets, and only authorized personnel could access this information. Data will be stored for up to 10 years.

Statistical analysis will be performed using the SPSS (SPSS Inc. Chicago, IL, USA). Data will be presented by percentage, mean and standard deviation, and median where appropriate. Chi-square test, Fisher's exact test, student-t test will be used for data analysis where appropriate. A two-tailed probability value of p< 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IUI cycles
* Infertility patients aged >18 years old and < 42 years old
* BMI <30 kg/m2
* No sexually transmitted diseases, AIDS, syphilis and other infectious disease

Exclusion Criteria:

* Concurrent administration of other agents such as prednisolone, intravenous immunoglobulin, or G-CSF
* Administration of anticoagulants or NSAIDs at least 7 days before PRP infuse
* Drug addiction
* Urinary tract infection
* Underlying uncontrolled diabetes or hypertension, chromosomal or uterine abnormalities, genetic, hematologic, immunological, or endocrine disorders
* Chronic disease, systemic disease or cancers
* Blood diseases (sepsis, thrombocytopenia)
* Haemoglobin < 11g/dL, platelet count < 150000 mm3
* Poor sperm samples (raw sample TMS <5 x 106)
* Smoking and drinking alcoholic beverages on the day of IUI
* Fever on the day of IUI

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | 6 weeks gestation and ultrasound scanning will be performed to confirm at least one gestational sac around 2 to 3 months after IUI.
  Rate of clinical pregnancy outcome in subjects undergoing IUI with PRP co-incubation with husband's sperm group than non-PRP group.

SECONDARY OUTCOMES:
Rate of potential infection or other complications | up to 24 weeks of IUI
  To evaluate the rate of potential infection or other complications such as ectopic pregnancy and molar pregnancy in the intervention group and control group
Sperm quality | up to 24 weeks of IUI
  Assessment of sperm quality Sperm quality will be assessed before raw semen, post isolated processed semen and after female PRP co-incubation with the processed semen

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pui Wah Chung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Obstetrics & Gynaecology The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided